CLINICAL TRIAL: NCT04503057
Title: Exhaled Breath Particles as a Clinical Indicator for Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS) in Coronavirus (Covid-19) Positive and Negative Patients
Brief Title: Exhaled Breath Particles as a Clinical Indicator for Lung Injury and Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PEx ARDS
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-01

CONDITIONS: Covid19; ARDS, Human; ALI
Keywords: Exhaled Breath Particles; Particles in Exhaled Air (PExA); COVID-19; ARDS; ALI
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood samples, broncho alveolar lavage sample, exhaled breath particles
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive: COVID-19-positive patients with pulmonary infection, ALI or ARDS
- COVID-19 negative: COVID-19-negative patients with pulmonary infection, ALI or ARDS

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) reflects the hallmark of the critical course of coronavirus (COVID19). The investigators have recently shown that Exhaled Breath Particles (EBP) measured as particle flow rate (PFR) from the airways could be used as a noninvasive real-time early detection method for primary graft dysfunction (which bears a pathophysiological resemblance to ARDS) in lung transplant patients. The investigators have also previously demonstrated the utility of PFR in early detection and monitoring of ARDS in a large animal model. PFR has been shown to be elevated prior to the cytokine storm which classically occurs in ARDS. Early detection of ALI and ARDS is intimately linked to a patient's chance of survival as early treatment consisting of the preparation for intensive care, prone positioning and protective mechanical ventilation can be implemented early in the process. In the present study the investigators aim to use real-time PFR as an early detector for COVID19-induced ARDS. The investigators will also collect EBPs onto a membrane for subsequent molecular analysis. Previous studies have shown that most of those proteins found in bronchoalveolar lavage (BAL) can also be detected in EBPs deposited on membranes. The investigators therefore also aim to be able to diagnose COVID19 by analyzing EBPs using Polymerase Chain Reaction (PCR) with the same specificity as PCR from BAL, with the added benefit of being able to identify protein biomarkers for early detection of ARDS.

DETAILED DESCRIPTION:
EBP will be measured on 100 patients who are coronavirus (COVID-19) positive as indicated by PCR tests. Measurement will be done on daily basis from the time the patient is admitted to the hospital as an inpatient until either discharge or transition to ICU care. The initiation of mechanical ventilation in ICU patients will facilitate the tracking of EBP patterns over the course of disease in each patient. EBP measurements will also be done on 100 patients without COVID19 infection who have normal lung function as a control cohort.

The study will involve measurements on patients who have been placed on mechanical ventilation in the ICU. The purpose of utilizing PFR will be to reduce the need for invasive diagnostic tests such as bronchoscopy and for hospital transportation associated with tests such as CT scans. This will ultimately serve to not only decrease the risk of infecting other patients and staff in the hospital environment, but also to facilitate careful monitoring of these critical patients by measuring the extent of lung injury over time. In addition to PFR, EBP will be collected and measured on a daily basis to track the EBP patterns on patients in mechanical ventilation. Pre-clinical studies have shown that EBP can measure the extent of lung injury over time (onset of ARDS and recovery (unpublished data))

Measurements are also planned for patients who are on mechanical ventilation on extracorporeal membrane oxygenation (ECMO) support as well.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALI
* Clinical diagnosis of ARDS
* COVID-19 infection as measured by a positive PCR test

Exclusion Criteria:

* Dementia
* Severe neurological disease
* Drug abuse

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary infection, ALI or ARDS. Patients on mechanical ventilation. Normal breathing patients. Patients on ECMO support.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of COVID-19 through PCR testing of EBPs | 12-36 months
  Real Time-PCR will be used to detect the presence of COVID-19 on membranes on which EBP have been collected to determine the efficacy of using the collection device for non-invasive detection of infection.
Protein concentration in EBP | 12-36 months
  Proteins will be measured in the samples of EBPs collected on the membrane for the purpose of identifying protein biomarkers of disease.
Particle flow rate (particles per minute) in exhaled air | 12-36 months
  The investigators have recently shown that Exhaled Breath Particles (EBP) measured as particle flow rate (PFR) from the airways could be used as a noninvasive real time early detection method for primary graft dysfunction (similar to ARDS) in lung transplant patients and for ARDS in a large animal model. PFR has been shown to increase before the cytokine storm which is a hallmark of ARDS. Early detection of ALI and ARDS is crucial for increasing a patient's chance of survival as it allows for early treatment, such as preparing for intensive care, prone positioning and protective mechanical ventilation settings. In the present study the investigators aim to use real-time PFR as an early detector for COVID-19-induced ARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt Ingemansson, MD, PhD, Principal Investigator — Region Skåne, Lund University
Locations (1):
- Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broberg E, Andreasson J, Fakhro M, Olin AC, Wagner D, Hyllen S, Lindstedt S. Mechanically ventilated patients exhibit decreased particle flow in exhaled breath as compared to normal breathing patients. ERJ Open Res. 2020 Feb 10;6(1):00198-2019. doi: 10.1183/23120541.00198-2019. eCollection 2020 Jan. PMID 32055633
- [Background] Stenlo M, Hyllen S, Silva IAN, Bolukbas DA, Pierre L, Hallgren O, Wagner DE, Lindstedt S. Increased particle flow rate from airways precedes clinical signs of ARDS in a porcine model of LPS-induced acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2020 Mar 1;318(3):L510-L517. doi: 10.1152/ajplung.00524.2019. Epub 2020 Jan 29. PMID 31994907
- [Background] Broberg E, Hyllen S, Algotsson L, Wagner DE, Lindstedt S. Particle Flow Profiles From the Airways Measured by PExA Differ in Lung Transplant Recipients Who Develop Primary Graft Dysfunction. Exp Clin Transplant. 2019 Dec;17(6):803-812. doi: 10.6002/ect.2019.0187. Epub 2019 Oct 11. PMID 31615381